CLINICAL TRIAL: NCT00550290
Title: Prophylactic Antibiotics for Prevention of Wound Complications Following Vulvectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2007.07.26.E2
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Wound Infection
Keywords: vulvectomy; wound infection; wound complication; prophylactic antibiotic; Post-operative wound complications following vulvectomy
MeSH Terms: conditions — Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Cefazolin Preoperatively (Active Comparator): Participants received Cefazolin 2 grams intravenously within 30 minutes prior to incision
  Interventions: Drug: Cefazolin Preoperatively
- Cefazolin Postoperatively (Experimental): Participants received Cefazolin 2 gram intravenous within 30 minutes prior to incision and 1 gram Cefazolin every 8 hours for the first 24 hours post-op
  Interventions: Drug: Cefazolin PostOperatively

INTERVENTIONS:
Drug: Cefazolin PostOperatively — Cefazolin 1 gram IV every 8 hours for a total of 3 doses. Patients in both arms will receive an initial pre-operative 2 gram dose of Cefazolin within 30 minutes prior to incision. In penicillin/cephalosporin allergic patients, the substitute of Clindamycin 900 mg IV q 8 hrs will be used.
  Other Names: Ancef; Kefzol
  Arms: Cefazolin Postoperatively
Drug: Cefazolin Preoperatively — Patients in active comparator arm will receive an initial pre-operative 2 gram does of Cefazolin within 30 minutes prior to incision. In penicillin/cephalosporin allergic patients, the substitute of Clindamycin 900 mg IV will be used.
  Other Names: Ancef; Kefzol
  Arms: Cefazolin Preoperatively

SUMMARY:
This randomized prospective study will specifically investigate the efficacy of a 24 hour post-operative course of broad-spectrum prophylactic antibiotics - namely Cefazolin - in preventing wound infection and wound breakdown following vulvectomy.

DETAILED DESCRIPTION:
Infectious morbidity in gynecologic oncology has not been thoroughly investigated to date. Included in the literature are several studies that highlight substantial numbers of post-surgical infectious complications. Specifically among patients undergoing radical vulvectomy, the incidence of post-operative wound complication is as high as 58%. Surgery is the treatment of choice for vulvar cancer, but few studies establish protocols or management strategies to prevent the complications of post-operative wound infection and breakdown. This proposed randomized prospective study would specifically investigate the efficacy of a 24 hour post-operative course of broad-spectrum prophylactic antibiotics - namely Cefazolin - in preventing wound infection and wound breakdown following vulvectomy. This same regimen has been described by a leader in the field of gynecology in his text - TeLinde's Operative Gynecology. This study will utilize two arms - one as the treatment arm utilizing 24 hours of prophylactic antibiotics and the other as control.

ELIGIBILITY:
Inclusion Criteria:

* All female patients 18 years of age or older undergoing surgery for vulvar carcinoma (this includes female patients undergoing any form of vulvectomy - radical, vulvectomy without groin node dissection, and partial vulvectomy)
* Disease State will not affect inclusion in the study. Women with previous surgery for vulvar carcinoma will be included as will those undergoing initial operation.
* Number of subjects: 160

Exclusion Criteria:

* Women simultaneously undergoing treatment for other forms of cancer
* Women under the age of 18
* Pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Hopkins, MD, Study Chair — Aultman Health Foundation; William T. Schnettler, MD, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Health Foundation, Canton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July, 2007 through December, 2008, all patients undergoing surgical treatment for vulvar cancer at a single tertiary care center were offered enrollment and randomization.
Groups:
- 24 Hour Post-operative Course of Cefazolin: Patients undergoing surgical treatment for vulvar cancer randomized to an extended 24 hour post-operative course of Cefazolin
- Pre-operative Single Dose of Cefazolin.: Patients randomized to the standard pre-operative single dosing regimen of Cefazolin.
Period: Overall Study
Arm/Group | 24 Hour Post-operative Course of Cefazolin | Pre-operative Single Dose of Cefazolin.
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24 Hour Post-operative Course of Cefazolin | Pre-operative Single Dose of Cefazolin. | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Wound Complications
Description: Number of participants experiencing wound complications following vulvectomy. The presence of febrile episodes, elevated WBC counts and exam findings will be used to diagnose wound complications.
Time Frame: Two-week post-operative
Population: All participants who received their assigned dose of each intervention and completed all study visits were included in the efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 24 Hour Post-operative Course of Cefazolin | Pre-operative Single Dose of Cefazolin.
Number analyzed (Participants) | 10 | 8
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | 24 Hour Post-operative Course of Cefazolin | Pre-operative Single Dose of Cefazolin.
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
Small number of subjects recruited lead to unreliable data. A larger sample is needed to answer the research question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No